CLINICAL TRIAL: NCT07158788
Title: Incremental Value of Frailty Indices in Bleeding Risk Prediction Among Patients With Acute Coronary Syndrome
Brief Title: Role of Frailty in Bleeding Risk Prediction in Acute Coronary Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mario Hosny Labib Habib, Resident physician, Assiut University
Other Study IDs: Frailty Bleeding ACS
Record Dates: First submitted 2025-09-04; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Frailty; Acute Coronary Syndrome; Bleeding
Keywords: Frailty; acute coronary syndrome; bleeding; bleeding risk prediction
MeSH Terms: conditions — Frailty; Acute Coronary Syndrome; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Studying the incremental role of frailty in predicting in-hospital, short-term (30 days), and mid-term (6 months) bleeding in ACS patients.

DETAILED DESCRIPTION:
Potent platelet inhibition reduces the risk of thrombotic complications in patients with acute coronary syndromes. Unavoidably, the more potent platelet inhibition increases the risk of bleeding. Bleeding risk can be predicted using the ARC-HBR criteria, the CRUSADE score, ACUITY score, and PRECISE-DAPT score. These conventional risk scores incorporate clinical, laboratory and procedural variables but often overlook patient centered geriatric parameters such as frailty. Frailty is a multidimensional syndrome characterized by decreased reserves and diminished resistance to stressors. It can be assessed using Rockwoods clinical frailty scale, the frailty index, frailty domains and the Fried scale. The association between frailty and bleeding risk in ACS patients is still inadequately studied. We hypothesize that frailty indices would increase the discriminatory power of established standard bleeding risk scores, and would predict bleeding events among ACS patients.

ELIGIBILITY:
Inclusion Criteria:

1. - Patients must be suffering from acute coronary syndrome ( STEMI - NSTEMI ) at the time of recruitment
2. - Patients must be older than 65 years

Exclusion Criteria:

1. - Patients younger than 65 years
2. - Refusal of participation
3. - In - hospital death unrelated to bleeding

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients presenting with acute coronary syndrome ( STEMI and NSTEMI) and are older than 65 years
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Bleeding Academic Research Consortium ( BARC ) type 3 to 5 | Baseline
  Type 3: Major bleeding (with subtypes) 3a: Overt bleeding plus hemoglobin drop of 3-5 g/dL, or Transfusion with ≤2 units of blood.
  3b: Hemoglobin drop ≥5 g/dL, Cardiac tamponade, Bleeding requiring surgical intervention, or Bleeding requiring intravenous vasoactive agents. 3c: Intracranial hemorrhage (excluding microbleeds), Intraocular bleeding compromising vision.
  Type 4: CABG-related bleeding Perioperative bleeding within 48 hours of coronary artery bypass grafting (CABG) and Reoperation for bleeding, ≥5 units of blood transfused, Chest tube output ≥2 L in 24 hours, or Cardiac tamponade.
  Type 5: Fatal bleeding 5a: Probable fatal bleeding (no autopsy or imaging confirmation). 5b: Definite fatal bleeding (confirmed by autopsy or imaging)

SECONDARY OUTCOMES:
Bleeding Academic Research Consortium ( BARC ) type 0, 1 or 2 | Baseline
  Type 0 : no bleeding Type 1: Bleeding that is not actionable and does not require medical attention Type 2 : Any bleeding that requires medical attention, hospitalization, or evaluation by a health care professional. but does not meet criteria for type 3, 4 or 5.